CLINICAL TRIAL: NCT06039345
Title: The Effectiveness of Shoulder Terminal Sensory Articular Nerve Radiofrequency Ablation for Non-surgical Refractory Shoulder Pain Due to Rotator Cuff Pathology and Osteoarthritis; A Prospective Pilot Study
Brief Title: Shoulder RFA Pilot Study
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Allison Glinka Przybysz, Assistant Professor, University of Utah
Other Study IDs: 159158
Record Dates: First submitted 2023-08-29; First posted 2023-09-15 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Pain; Rotator Cuff Injuries
Keywords: shoulder radiofrequency ablation
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through this prospective, single-arm cohort pilot study, we plan to explore the safety and effectiveness of Shoulder Radiofrequency Ablation (SRFA) in patients with non-operative chronic shoulder pain due to shoulder osteoarthritis with or without rotator cuff tears.

DETAILED DESCRIPTION:
This will be one of the first collaborative prospective, single-arm cohort using a standardized selection protocol and comprehensive SRFA protocol to treat chronic, refractory shoulder pain due radiographically confirmed glenohumeral joint OA with or without RTC pain, in patients deemed non-surgical candidates by a board-certified orthopedic shoulder surgeon. Upon completing the proposed research, we expect our contribution to fill the knowledge gap on whether SRFA is a potentially viable treatment option for this patient population. This contribution is expected to be substantial because SRFA may be a safe and effective treatment option for many people suffering shoulder pain and debility who are sub-optimal surgical candidates and have historically either been undertreated to have less than ideal treatments options, including opioid-based pain management in particular.

ELIGIBILITY:
Inclusion Criteria:

1. ≥50 years old capable of understanding and providing consent in English, and capable of complying with the outcome instruments used
2. ≥3 months of shoulder pain refractory to conventional treatment (i.e., physiotherapy, medication, steroid injections)
3. Persistent shoulder pain ≥ 4/10 in intensity on a 7-day average
4. Shoulder pain refractory to conventional treatment (i.e., physical therapy, oral analgesics, steroid injection)
5. Prior consultation with a board-certified orthopedic shoulder surgeon, deemed a non-surgical candidate for the primary diagnosis of glenohumeral joint pain +/- rotator cuff pain
6. ≥80% pain relief for at least 30 minutes after a single fluoroscopically-guided block of the sensory branches of the SN, AN, and LPN with 0.5 mL of lidocaine at each nerve
7. Scheduled for procedure of interest

Exclusion Criteria:

1. Infection
2. Allergy to any medication needed to participate in this study
3. Previous partial/total/reverse shoulder arthroplasty. Participants with a history of RTC repair will not be excluded.
4. Neurologic disorders including radiculopathy, connective tissue/inflammatory joint disease/widespread soft tissue pain disorder
5. Severe, uncontrolled psychiatric disorder requiring hospitalization within 6 months
6. Intraarticular or subacromial injection to the study shoulder within 3 months before C-SRFA
7. Uncontrolled bleeding diathesis
8. Pregnancy
9. Pacemaker, neurostimulator, or other implanted device potentially sensitive to RF energy
10. Active Worker's compensation claim, litigation, or other possible reason for secondary gain.
11. Prior shoulder radiofrequency ablation
12. Daily opioid use

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will explore the effectiveness of SRFA to reduce chronic shoulder pain in 10 participants who were deemed non-surgical candidates by an orthopedic surgeon and who experienced ≥80% pain relief after a single shoulder joint anesthetic block.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) at 1, 3, 6 and 12 months after the SRFA | 1, 3, 6 and 12 months
  Pain reduction will be measured by calculating the proportion of participants who experienced ≥50% reduction of their shoulder pain on the Numerical Rating Scale (NRS) at 1, 3, 6 and 12 months after the SRFA.

SECONDARY OUTCOMES:
Myotomal strength at 1, 3, 6 and 12 months after SRFA | 1, 3, 6 and 12 months after SRFA
  We will calculate the proportion of participants who experience a minimal clinically important difference (MCID) in shoulder abduction, elbow flexion, wrist extension, elbow extension and hand grip measured by dynamometer after SRFA. We will do this by calculating the proportion of participants who experience ≥20% change (MCID) in myotomal strength at 1, 3, 6 and 12 months after SRFA.
American Shoulder and Elbow Surgeons Score (ASES) at 1,3, 6 and 12 months after SRFA | 1, 3, 6 and 12 months after SRFA
  We will use the validated American Shoulder and Elbow Surgeons Score (ASES) questionnaire to calculate the proportion of participants who experience an MCID on ASES (defined as a score of ≥ 7) at 1,3, 6 and 12 months after SRFA.
Patient Global Impression of Change (PGIC) at 1,3, 6 and 12 months after SRFA | 1, 3, 6 and 12 months after SRFA
  We will use the validated Patient Global Impression of Change (PGIC) questionnaire to calculate the proportion of participants who experience an MCID on PGIC (defined as a score of ≥ 5) at 1,3, 6 and 12 months after SRFA.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Utah Farmington Health Center, Farmington, Utah
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - University of Utah South Jordan Health Center, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson HI, Ejlertsson G, Leden I, Rosenberg C. Chronic pain in a geographically defined general population: studies of differences in age, gender, social class, and pain localization. Clin J Pain. 1993 Sep;9(3):174-82. doi: 10.1097/00002508-199309000-00004. PMID 8219517
- [Background] Chard MD, Hazleman R, Hazleman BL, King RH, Reiss BB. Shoulder disorders in the elderly: a community survey. Arthritis Rheum. 1991 Jun;34(6):766-9. doi: 10.1002/art.1780340619. PMID 2053923
- [Background] Allander E. Prevalence, incidence, and remission rates of some common rheumatic diseases or syndromes. Scand J Rheumatol. 1974;3(3):145-53. doi: 10.3109/03009747409097141. No abstract available. PMID 4428194
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Virta L, Joranger P, Brox JI, Eriksson R. Costs of shoulder pain and resource use in primary health care: a cost-of-illness study in Sweden. BMC Musculoskelet Disord. 2012 Feb 10;13:17. doi: 10.1186/1471-2474-13-17. PMID 22325050
- [Background] Eckmann MS, Bickelhaupt B, Fehl J, Benfield JA, Curley J, Rahimi O, Nagpal AS. Cadaveric Study of the Articular Branches of the Shoulder Joint. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):564-570. doi: 10.1097/AAP.0000000000000652. PMID 28786899
- [Background] Eckmann MS, Johal J, Bickelhaupt B, McCormick Z, Abdallah RT, Menzies R, Soliman S, Nagpal AS. Terminal Sensory Articular Nerve Radiofrequency Ablation for the Treatment of Chronic Intractable Shoulder Pain: A Novel Technique and Case Series. Pain Med. 2020 Apr 1;21(4):868-871. doi: 10.1093/pm/pnz335. No abstract available. PMID 31851366
- [Background] Bohannon RW. Reference values for extremity muscle strength obtained by hand-held dynamometry from adults aged 20 to 79 years. Arch Phys Med Rehabil. 1997 Jan;78(1):26-32. doi: 10.1016/s0003-9993(97)90005-8. PMID 9014953
- [Background] Bohannon RW. Grip strength impairments among older adults receiving physical therapy in a home-care setting. Percept Mot Skills. 2010 Dec;111(3):761-4. doi: 10.2466/03.10.15.PMS.111.6.761-764. PMID 21319615
- [Background] Hayes K, Walton JR, Szomor ZL, Murrell GA. Reliability of 3 methods for assessing shoulder strength. J Shoulder Elbow Surg. 2002 Jan-Feb;11(1):33-9. doi: 10.1067/mse.2002.119852. PMID 11845146
- [Background] Kolber MJ, Beekhuizen K, Cheng MS, Fiebert IM. The reliability of hand-held dynamometry in measuring isometric strength of the shoulder internal and external rotator musculature using a stabilization device. Physiother Theory Pract. 2007 Mar-Apr;23(2):119-24. doi: 10.1080/09593980701213032. PMID 17530541
- [Background] Awatani T, Mori S, Shinohara J, Koshiba H, Nariai M, Tatsumi Y, Nagata A, Morikita I. Same-session and between-day intra-rater reliability of hand-held dynamometer measurements of isometric shoulder extensor strength. J Phys Ther Sci. 2016 Mar;28(3):936-9. doi: 10.1589/jpts.28.936. Epub 2016 Mar 31. PMID 27134388
- [Background] Michener LA, McClure PW, Sennett BJ. American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section: reliability, validity, and responsiveness. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):587-94. doi: 10.1067/mse.2002.127096. PMID 12469084
- [Background] Jones IA, Togashi R, Heckmann N, Vangsness CT Jr. Minimal clinically important difference (MCID) for patient-reported shoulder outcomes. J Shoulder Elbow Surg. 2020 Jul;29(7):1484-1492. doi: 10.1016/j.jse.2019.12.033. Epub 2020 Apr 3. PMID 32249146
- [Background] Conger A, Gililland J, Anderson L, Pelt CE, Peters C, McCormick ZL. Genicular Nerve Radiofrequency Ablation for the Treatment of Painful Knee Osteoarthritis: Current Evidence and Future Directions. Pain Med. 2021 Jul 25;22(Suppl 1):S20-S23. doi: 10.1093/pm/pnab129. PMID 34308957
- [Background] Conger A, Cushman DM, Walker K, Petersen R, Walega DR, Kendall R, McCormick ZL. A Novel Technical Protocol for Improved Capture of the Genicular Nerves by Radiofrequency Ablation. Pain Med. 2019 Nov 1;20(11):2208-2212. doi: 10.1093/pm/pnz124. PMID 31131850
- [Background] Koshi E, Cheney CW, Sperry BP, Conger A, McCormick ZL. Genicular Nerve Radiofrequency Ablation for Chronic Knee Pain Using a Three-Tined Electrode: A Technical Description and Case Series. Pain Med. 2020 Dec 25;21(12):3344-3349. doi: 10.1093/pm/pnaa204. PMID 32984887
- [Background] McCormick ZL, Cohen SP, Walega DR, Kohan L. Technical considerations for genicular nerve radiofrequency ablation: optimizing outcomes. Reg Anesth Pain Med. 2021 Jun;46(6):518-523. doi: 10.1136/rapm-2020-102117. Epub 2021 Jan 22. PMID 33483425
- [Background] McCormick ZL, Reddy R, Korn M, Dayanim D, Syed RH, Bhave M, Zhukalin M, Choxi S, Ebrahimi A, Kendall MC, McCarthy RJ, Khan D, Nagpal G, Bouffard K, Walega DR. A Prospective Randomized Trial of Prognostic Genicular Nerve Blocks to Determine the Predictive Value for the Outcome of Cooled Radiofrequency Ablation for Chronic Knee Pain Due to Osteoarthritis. Pain Med. 2018 Aug 1;19(8):1628-1638. doi: 10.1093/pm/pnx286. PMID 29300971
- [Background] Roberts SL, Stout A, Dreyfuss P. Review of Knee Joint Innervation: Implications for Diagnostic Blocks and Radiofrequency Ablation. Pain Med. 2020 May 1;21(5):922-938. doi: 10.1093/pm/pnz189. PMID 31407791
- [Background] Tran A, Reiter DA, Fritz J, Cruz AR, Reimer NB, Lamplot JD, Gonzalez FM. Pilot study for treatment of symptomatic shoulder arthritis utilizing cooled radiofrequency ablation: a novel technique. Skeletal Radiol. 2022 Aug;51(8):1563-1570. doi: 10.1007/s00256-022-03993-y. Epub 2022 Jan 14. PMID 35029737
- [Background] Eckmann MS, McCormick ZL, Beal C, Julia J, Cheney CW, Nagpal AS. Putting Our Shoulder to the Wheel: Current Understanding and Gaps in Nerve Ablation for Chronic Shoulder Pain. Pain Med. 2021 Jul 25;22(Suppl 1):S2-S8. doi: 10.1093/pm/pnab152. PMID 34308959
- [Background] Bogduk N. On diagnostic blocks for lumbar zygapophysial joint pain. F1000 Med Rep. 2010 Aug 9;2:57. doi: 10.3410/M2-57. PMID 21173871
- [Background] Schneider BJ, Joshi M, Ehsanian R, McCormick ZL, Patel J, Zheng P, Nagpal AS. Patient-perceived duration of effect of lidocaine and bupivacaine following diagnostic medial branch blocks; a multicenter study. Interv Pain Med. 2022 Mar 18;1(2):100083. doi: 10.1016/j.inpm.2022.100083. eCollection 2022 Jun. PMID 39239364
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Diagnosis and treatment of incomplete rotator cuff tears - PubMed. Accessed June 22, 2022. https://pubmed.ncbi.nlm.nih.gov/2182260/